CLINICAL TRIAL: NCT02981706
Title: A Pilot Randomized Trial of Arteriovenous Fistula (AVF) Versus Arteriovenous Graft (AVG) in Elderly Patients With Advanced Chronic Kidney Disease (CKD)
Brief Title: Comparison of AVF Versus AVG in Elderly Patients Starting Dialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Maya Rao, Assistant Professor of Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAQ8223; R03AG053294 (NIH)
Record Dates: First submitted 2016-11-30; First posted 2016-12-05 (Estimated); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Chronic Kidney Disease; Endstage Renal Disease
Keywords: Arteriovenous Fistula (AVF); Arteriovenous Graft (AVG)
MeSH Terms: conditions — Renal Insufficiency, Chronic; Arteriovenous Fistula | interventions — Arteriovenous Shunt, Surgical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arteriovenous Fistula (AVF) Group (Active Comparator): Patient will receive an arteriovenous fistula (connection between native artery and vein) as his/her dialysis access
  Interventions: Procedure: Arteriovenous Fistula (AVF)
- Arteriovenous Graft (AVG) Group (Active Comparator): Patient will receive an arteriovenous graft (synthetic connection between artery and vein) as his/her dialysis access
  Interventions: Procedure: Arteriovenous Graft (AVG)

INTERVENTIONS:
Procedure: Arteriovenous Fistula (AVF) — The location of vascular access placement in the upper extremity will be based on pre-surgery vein mapping and the appearance of the vessels at the time of the surgery, with the most distal clinically acceptable location used. When no contra-indication is present, the vascular access will be placed in the non-dominant arm per standard of care. In this case, the vascular access will be an arteriovenous fistula, or connection between a native artery and vein.
  Other Names: AVF
  Arms: Arteriovenous Fistula (AVF) Group
Procedure: Arteriovenous Graft (AVG) — The location of vascular access placement in the upper extremity will be based on pre-surgery vein mapping and the appearance of the vessels at the time of the surgery, with the most distal clinically acceptable location used. When no contra-indication is present, the vascular access will be placed in the non-dominant arm per standard of care. In this case, the vascular access will be an arteriovenous graft, or synthetic connection between a native artery and vein.
  Other Names: AVG
  Arms: Arteriovenous Graft (AVG) Group

SUMMARY:
This is a pilot, single-center, randomized trial of 90 subjects to evaluate complication rates and functional status decline in subjects age 65 years and older referred for vascular access placement. Subjects will be randomized to arteriovenous fistula (AVF) (n = 45) versus arteriovenous graft (AVG) (n = 45), placed in a vascular access monitoring protocol, and undergo measurements of functional status including gait speed, grip strength, and self-reported function over 6 months. The primary hypothesis to be tested is that AVF placement will result in a higher proportion of primary access failure as defined by a binary composite primary endpoint of an unsalvageable access or an immature access or a non-functional access measured at 6 months compared to AVG placement. In addition, the study will evaluate whether AVF placement and a greater number of access procedures will result in a greater decline in functional status as measured by the average change over 6 months in gait speed, grip strength, and self-reported function as assessed by the Disabilities in Arm, Shoulder and Hand Survey.

DETAILED DESCRIPTION:
The elderly population is the fastest growing segment of the dialysis population. A vascular access is required to perform dialysis and current guidelines support arteriovenous fistulas (AVFs) over arteriovenous grafts (AVGs) as the preferred vascular access for dialysis. However, the preferred choice of vascular access in the elderly is unclear. Older adults have higher rates of complications from AVF placement compared to AVG placement. Placement of a dialysis access and the procedures subsequently required to achieve and maintain access functionality could result in further declines of function in this already frail population and potentially reduce quality of life. High burdens of cardiovascular disease, heterogeneous life expectancy and variable health goals may make the ideal choice of vascular access different in the elderly population than the general dialysis population.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years or older
* Referred by nephrology provider for vascular access for hemodialysis (HD)
* Able and willing to provide informed consent

Exclusion Criteria:

* Patient is not a candidate for an AVF per surgeon
* Congestive heart failure (CHF) as defined by ejection fraction (EF) < 20%, history of heart transplant, history of ventricular assist device
* Known central venous stenosis
* Metastatic cancer or active cancer receiving chemotherapy
* Multiple Myeloma
* Vein mapping with arterial diameter ≤ 2mm and vein diameter ≤ 2.5mm or presence of stenosis or thrombosis in the draining vein
* arterial flow velocity of ≤ 40ml/min

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-10-06 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
Proportion of Patients with Primary Access Failure | Up to 6 months after procedure
  Primary access failure as defined by a binary composite primary endpoint of an unsalvageable access or an immature access or a non-functional access measured at 6 months.
  An access determined to be unsalvageable by the vascular surgeon and requiring a new access placement will meet the primary endpoint. For subjects on HD at 6 months, self-report of successful use of the vascular access three times will be considered functional and will not meet the primary endpoint. For all subjects not on HD at 6 months, ultrasound will be performed and interpreted by the vascular surgeon, and a mature, functioning access will be defined as meeting the following criteria:1) 600ml/min blood flow, 2) 6mm diameter dilation of the access, and 3) 6mm or less depth from the skin to the access. Any vascular access that does not fulfill all three criteria will meet the primary endpoint.

SECONDARY OUTCOMES:
Mean Number of Procedures Between the Two Groups | Up to 6 months after the procedure
  The number of surgical and endovascular procedures after the initial vascular access placement measured at 6 months.
Time to Event | Up to 6 months after the procedure
  A time to event analysis will be performed looking at the time to successful use of the vascular access. This will be defined either as self-report of being used at dialysis three times successfully or an ultrasound showing a mature, functioning access defined as meeting the following criteria: 1) 600ml/min blood flow, 2) 6mm diameter dilation of the access, and 3) 6mm or less depth from the skin to the access.
Change in Gait Speed | Baseline, 3 months, 6 months
  The average decline in meters/second between subjects who receive AVF versus AVG and also subjects who have < 2 versus ≥ 2 number of access procedures after the initial access placement.
Change in Grip Strength | Baseline, 3 months, 6 months
  Compare the average decline in kilograms between subjects who receive AVF versus AVG and also subjects who have < 2 versus ≥ 2 number of access procedures after the initial access placement. In addition, for each subject we will measure the difference in grip strength from time zero to 6 months between the ipsilateral hand and contralateral hand from the access placement. We will compare the mean grip strength difference between the ipsilateral and contralateral hand between the AVF and AVG group using a two-sample t-test.
Change in Disabilities of the Arm, Shoulder and Hand (DASH) Score | Baseline, 3 months, 6 months
  Compare the mean change in score from 0 - 100 between subjects who receive AVF versus AVG and also subjects who have < 2 versus ≥ 2 number of access procedures after the initial access placement.
  The DASH Outcome Measure is scored in two components: the disability/symptom section (30 items, scored 1-5) and the optional high performance Sport/Music or Work section (4 items, scored 1-5). For this study, we will only use to the disability/symptom section score.
Change in Cognitive Screen | Baseline and 6 months
  The difference between the number of people who go from a negative to a positive screen between the two groups (AVF vs AVG and < 2 versus ≥ 2 number of access procedures).

CONTACTS AND LOCATIONS:
Overall Officials: Maya Rao, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Data will be retained by the Columbia PI for future research use. This applies only to those subjects who consent to allow the storage and use of their data in identifiable form after completion of the study